CLINICAL TRIAL: NCT02638415
Title: The Effect of HVPG-Guided Individualized Therapy in Patients With Cirrhosis Related Esophagogastric Variceal Hemorrhage For Secondary Prophylaxis:A Randomized Controlled Trial
Brief Title: The Effect of Hepatic Vein Pressure Gradient(HVPG)-Guided Therapy in Cirrhotic Patients With Esophagogastric Varices
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Public Health Clinical Center (Other Government); ShuGuang Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Pudong New Area Gongli Hospital (Other); Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, Director of department of Gastroenterology, Zhongshan Hospital, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSY-WYC02-2015
Record Dates: First submitted 2015-12-09; First posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Gastroesophageal Varices; Cirrhosis
Keywords: HVPG
MeSH Terms: conditions — Fibrosis | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HVPG group (Experimental): HVPG-guided therapy
  Interventions: Procedure: HVPG-guided therapy; Drug: Carvedilol
- non-HVPG group (Other): routine therapy
  Interventions: Other: routine therapy; Drug: Carvedilol

INTERVENTIONS:
Procedure: HVPG-guided therapy — Patients with an HVPG over 20mmHg will be suggested to receive transjugular intrahepatic portocaval shunt (TIPS) or surgical shunt operation.
  Patients with an HVPG between 16 and 20mmHg can choose either endoscopic treatment or TIPS according their willingness and indication.
  Patients with an HVPG below 16mmHg will be treated by endoscopy plus Carvedilol, until endoscopic treatment fails.
  Arms: HVPG group
Other: routine therapy — Patients start treatment without HVPG measurement and receive endoscopic therapy plus Carvedilol.
  Arms: non-HVPG group
Drug: Carvedilol — Patients in HVPG group with HVPG below 16mmHg and all patients in non-HVPG group will take Carvedilol 12.5mg/d if they have no contraindications.

SUMMARY:
The purpose of the study is to compare the effect of HVPG-guided individualized therapy and non-HVPG guided traditional therapy in cirrhotic patients for secondary prophylaxis.

DETAILED DESCRIPTION:
The study is a randomized controlled trial of Zelen-design. Patients randomly enter two treatment groups: 1) the HVPG group and 2) the non-HVPG group. Treatment allocation is by block randomization with an equal number for both groups. The results are concealed in opaque envelopes.After randomization, patients will have a second chance to decide if they want to stay in the current group.Patients can switch to another group according to their will. If they are in the HVPG group，they will receive HVPG measurement before treatment. If they are in the non-HVPG group, they start treatment without HVPG measurement and receive endoscopic treatment plus Carvedilol.The mortality rate and rebleeding rate will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis diagnosed by histology, radiological evidence of cirrhosis, and endoscopic evidence of varices;
* Patients with a previous history of variceal hemorrhage;
* Patients admitted to Zhongshan Hospital and other 6 tertiary centers in Shanghai from Dec 1, 2015 to Sep 31,2018

Exclusion Criteria:

* Patients already taken secondary prophylactic treatment including endoscopic, pharmacological, surgical and interventional therapies;
* Patients with severe systemic diseases such as chronic heart failure or chronic renal failure that will have impact on survival;
* Patients in pregnancy and lactation;
* Patients already diagnosed with hepatic cellular carcinoma or other malignant tumors;
* Patients with contraindication to treatment of endoscopy, surgery and TIPS: severe coagulation defects, allergic to contrast medium used in TIPS, hepatic encephalopathy, spontaneous bacterial peritonitis;
* Patients with conditions that will influence the accuracy of HVPG measurement: Cavernous transformation of portal vein, diffused portal vein thrombosis, severe shunt;
* Patients refuse to give consent to the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | through study completion, an average of 1 year
  The investigators observe the mortality events in both groups during the study

SECONDARY OUTCOMES:
Rebleeding rate | through study completion, an average of 1 year
  The investigators observe the rebleeding events in both groups during the study
Adverse Events | through study completion, an average of 1 year
  The investigators observe any severe adverse events caused by HVPG measurement, endoscopic procedures,use of Carvedilol, surgical operations or TIPS
Total cost | through study completion, an average of 1 year
  The investigators calculate the total cost of treatment of each patient during the study

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, Professor, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China